CLINICAL TRIAL: NCT01381042
Title: Retrospective Study on the Incidence and Factors of Brown Adipose Tissue in Adult Chinese
Brief Title: The Incidence and Factors of Brown Adipose Tissue in Chinese
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Yiming Li, Division of Endocrinology and Metabolism
Other Study IDs: KY2009-307
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2009-12

CONDITIONS: Obesity
Keywords: Brown Adipose Tissue; Incidence; Factor; Human
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Previous studies have shown active brown adipose tissue (BAT) is present in adults and may play important roles in regulating energy homeostasis. However, the majorities of these studies were done in patients undergoing scanning for cancer surveillance, and may not reflect BAT behavior in healthy individuals. In addition, little is known about the ethnic variation in BAT activity, particularly in Chinese adults. Due to the large amount in our cohort, we are able to look at the difference between subjects for cancer surveillance (CS) and subjects for medical check-up (MC), and to clarify the impact of clinical and lifestyle parameters.

DETAILED DESCRIPTION:
We will study scanning database including data from July 2006 to June 2010 in Shanghai. BAT activity will be measured via 18F-fluorodeoxyglucose (FDG) positron emission tomography/computed tomography (PET/CT). Age, imaging date, sex, and outdoor temperature will be collected for all patients. To evaluate the effects of multiple metabolic parameters on BAT activity, we will collect height, body weight, fasting plasma glucose (FPG), medical history, diagnosis, smoking, alcohol consumption, exercise, liver triglyceride content, and thyroid metabolic activity for all patients with detectable BAT and their negative controls, consisting of two patients who underwent PET/CT scans at the same day but without detectable BAT.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with detectable brown adipose tissue
* Negative controls, consisting of two subjects who underwent PET/CT scans at the same day but without detectable BAT

Exclusion Criteria:

* Younger than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who underwent scanning for either cancer surveillance (CS) or medical check-up (MC) from July 2006 to June 2010 in Huashan Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yiming Li, Dr., Study Chair — Huashan Hospital
Locations (1):
- Huashan Hospital, Shanghai, China